CLINICAL TRIAL: NCT04520698
Title: Utilizing Palliative Leaders In Facilities to Transform Care for Alzheimer's Disease
Acronym: UPLIFT-AD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: University of Maryland, Baltimore (Other); National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Kathleen T. Unroe, Associate Professor of Medicine, Indiana University
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: 2005967061; R01AG066922 (NIH)
Record Dates: First submitted 2020-08-17; First posted 2020-08-20 (Actual); Last update posted 2025-10-23 (Actual); Status verified 2025-10

CONDITIONS: Alzheimer Disease
Keywords: Alzheimer Disease; Palliative Care; Dementia; Nursing Home
MeSH Terms: conditions — Alzheimer Disease; Dementia

STUDY DESIGN:
Intervention Model Description: The study will use a stepped-wedge non-randomized trial design with 16 sites in two states (Indiana and Maryland). The study team will compare process and outcomes of the UPLIFT-AD intervention vs. usual care. The intervention will be implemented consecutively over 36 months, with staggered roll-out at 4 sites (2 per state) approximately every 6 months.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Nursing Home-level UPLIFT-AD intervention (Experimental): The UPLIFT-AD intervention consists of three major components delivered at the level of the nursing home: 1) in-house PC champions trained to a) facilitate advance care planning conversations with residents with Alzheimer's Disease and Related Dementias and their surrogate decision-makers, b) screen and follow up on residents' Palliative Care needs and c) serve as a liaison to Palliative Care consultants; 2) specialty Palliative Care consultant support providing individual consults for residents with complex Palliative Care needs; and 3) education on primary Palliative Care offered to all clinical NH staff.
  Interventions: Behavioral: UPLIFT-AD
- Usual Care (No Intervention): Usual nursing home care.

INTERVENTIONS:
Behavioral: UPLIFT-AD — Access to palliative care needs screening, advance care planning conversations, palliative care consultations
  Arms: Nursing Home-level UPLIFT-AD intervention

SUMMARY:
The purpose of this study is to evaluate a comprehensive model for integrating both primary and specialty Palliative Care for older adults with dementia into nursing facilities. Palliative Care is a supportive care approach that aims to improve the quality of life of patients and their families facing serious or life-threatening illnesses, through the prevention and relief of suffering through the treatment of pain and other problems, using physical, psychosocial and spiritual approaches. Palliative care is specialized medical care for people who are living with a serious illness. This type of care is focused on providing relief from the symptoms and from the stress of the illness. The goal is to improve quality of life for both patient and family.

The UPLIFT-AD model will include providing education on primary Palliative Care for residents with dementia to nursing facility staff, training nursing facility staff in providing primary Palliative Care, and providing access to specialty Palliative Care consultations for residents. To help understand the impact of these interventions, this study will also collect information about resident health, the care they receive, and perceptions of their quality of life according to both family members and nursing facility staff.

DETAILED DESCRIPTION:
The objective of this proposal is to evaluate the effectiveness of the UPLIFT-AD (Utilizing Palliative Leaders In Facilities to Transform care for Alzheimer's Disease) intervention and to assess the implementation context of the intervention using a hybrid 1 trial design. The UPLIFT-AD intervention includes 1) in-house PC champions trained to facilitate goals of care conversations with residents with Alzheimer's Disease and Related Dementias (ADRD) and their surrogate decision-makers, screen residents for symptoms and other PC needs, provide symptom management and serve as a liaison to external PC consultants; 2) specialty PC consultants who provide consults for complex residents and families; and 3) primary PC education for nursing home (NH) staff. The study will use a randomized, stepped wedge design involving 16 diverse NHs in Indiana and Maryland and 640 residents, 640 family members and/or surrogate decision-makers, and 320 nursing facility staff.

ELIGIBILITY:
Inclusion Criteria:

-

NURSING HOME RESIDENTS:

* Long-stay resident in an enrolled nursing home defined as not paying through Medicare Part A at the enrolled facility.
* Has a diagnosis of moderate to severe ADRD, as measured on the Minimum Data Set (MDS)
* Length of stay >30 days

FAMILY MEMBERS/SURROGATE DECISION MAKERS:

* Family member and/or surrogate decision maker for an eligible resident in an enrolled nursing home
* English-speaking

NURSING HOME STAFF:

* Staff, nurse, or nurse assistant in an enrolled nursing facility
* English-speaking

Exclusion Criteria:

-

NURSING HOME RESIDENTS:

• Short-stay resident, defined as paying through Medicare Part A at the enrolled facility and/or receiving respite care

FAMILY MEMBERS/SURROGATE DECISION MAKERS:

• Non-English-speaking

NURSING FACILITY STAFF:

• Non-English-speaking

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1322 (Actual)
Dates: Start 2021-09-08 (Actual); Primary Completion 2025-09-30 (Actual); Study Completion 2025-09-30 (Actual)

PRIMARY OUTCOMES:
Change in End-of-Life Dementia - Comfort Assessment In Dying scale (EOLD-CAD) | Baseline (prior to intervention) and12 months (post intervention implementation)
  Nursing home staff and family members reported symptom frequency and intensity for 18 symptoms in the past 30 days. Symptom assessment was derived from the End-of-Life in Dementia Comfort Assessment in Dying (EOLD-CAD) and End-of-Life in Dementia Symptom Management (EOLD-SM) instruments. These symptoms included pain, discomfort, shortness of breath, choking, gurgling, difficulty swallowing, skin breakdown, restlessness, agitation, anxiety, depression, fear, crying, moaning, resistiveness to care, calm, serenity, peace. If the symptom did occur, respondents were asked if it had occurred once a month, 2-3 days a month, once a week, several days a week, or every day (ranging 0-5) and asked if the symptom was not at all intense, somewhat intense or very intense (ranging 1-3). Frequency and intensity were multiplied together for a score of 0-15 per symptom. A total score was derived by calculating the sum score and dividing by number of items. Higher scores indicate greater symptom burden.

SECONDARY OUTCOMES:
Change in End of Life Dementia - Satisfaction with Care (EOLD-SWC) scale | Baseline (prior to intervention) and 12 months (post intervention implementation)
  The outcome measure is change in the EOLD-SWC scale score. Participating family members/surrogate decisionmakers provided answers to questions asked over a 30 day timeframe. There are 10 items, each measured on a 4-point Likert scale ranging from 1 to 4 as follows: strongly disagree, disagree, agree, strongly agree. The items are added together for a cumulative score for a range of 10-40, with higher scores indicating greater satisfaction with care. The questionnaire items address decision-making, communication with health care professionals, understanding the resident's condition, and the resident's medical and nursing care.
Change in Quality-of-life (QOL) | Baseline (prior to intervention) and 12 months (post intervention implementation)
  The outcome measure is change in the quality-of-life (QOL) measure scale score. Two quality-of-life questions were asked of nursing home staff and family/surrogate decisionmakers about the respective resident's quality of life. One quality-of-life measure is a seven point scale describing overall quality of life. Another is a five point scale describing quality of life. Lower scores indicate poorer quality of life.
Change in staff palliative care knowledge | Baseline and 6 months (post intervention implementation)
  Change in staff palliative care knowledge will be measured by the Palliative Care survey (PCS). The PCS is a validated instrument, which includes subscales evaluating the frequency of key PC practice behaviors: family communication, provider coordination, planning/intervention, and bereavement. The total instrument score and each of the subscales are averaged to produce a range from 1 to 4, with higher scores indicating superior PC practices.
Quality of Dying in Long-Term Care (QOD-LTC) | Collected post-death
  The quality of dying-long-term care (QOD-LTC) scale was developed for cognitively impaired and intact residents. It was developed to be reported post-death for residents in NHs and residential care/assisted living settings. It assesses perspectives on quality of personhood, closure, and preparatory tasks. Higher mean scores reflect a higher quality of end-of-life in LTC. This was collected from nursing home staff and family/surrogate decisionmakers.
Change in Family Distress in Advanced Dementia Scale (Modified) | Baseline (prior to intervention) and 12 months (post intervention implementation)
  The Family Distress in Advanced Dementia Scale was developed for use with family members of nursing home residents with advanced dementia. Eighteen items from the scale were asked, consisting of three domains of distress: emotional distress, dementia preparedness, and nursing home relations . Higher scores indicate higher distress. Collected from family/surrogate decisionmakers only.

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen T Unroe, MD, MHA, Principal Investigator — Indiana University; John Cagle, PhD, MSW, Principal Investigator — University of Maryland, Baltimore
Locations (1):
- American Senior Communities, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: Yes
A de-identified dataset will be created for the purposes of sharing with qualified users, along with data content, format, and organization, will be stored at Indiana University and be available through the Co-PIs. Deidentified data will be available to qualified users who execute Data Use Agreements (DUAs) with the research team and NH partners.
Supporting Information: CSR, Analytic Code
Time Frame: The final de-identified dataset will be available to qualified investigators who meet the above criteria upon the on-line publication date of the final results of the trial.
Access Criteria: Individuals requesting access to the data must provide the following: (1) Executed DUAs with all NH partners; (2) documentation of Institutional Review Board approval; (3) a written commitment that the data will be used only for scholarly research purposes; (4) a written commitment that the user will not attempt to identify any individual patient or NH; (5) confirmation that the data will be secured using appropriate computer technology; and (6) a written commitment that data will be destroyed or returned after analyses are completed.

REFERENCES:
- [Derived] Unroe KT, Ersek M, Stump TE, Floyd A, Nesvet M, Block LVD, Tu W, Cagle JG. Discordance in Ratings of Symptoms Experienced by Nursing Home Residents With Cognitive Impairment. J Pain Symptom Manage. 2025 Nov 28:S0885-3924(25)00976-5. doi: 10.1016/j.jpainsymman.2025.11.022. Online ahead of print. PMID 41319818
- [Derived] Cagle JG, Stump TE, Tu W, Ersek M, Floyd A, Van den Block L, Zhang P, Becker TD, Unroe KT. A Psychometric Evaluation of the Staff-Reported EOLD-CAD Measure Among Nursing Home Residents With Cognitive Impairment. Int J Geriatr Psychiatry. 2025 Jan;40(1):e70037. doi: 10.1002/gps.70037. PMID 39743326
- [Derived] Unroe KT, Ersek M, Tu W, Floyd A, Becker T, Trimmer J, Lamie J, Cagle J. Using Palliative Leaders in Facilities to Transform Care for People with Alzheimer's Disease (UPLIFT-AD): protocol of a palliative care clinical trial in nursing homes. BMC Palliat Care. 2023 Jul 26;22(1):105. doi: 10.1186/s12904-023-01226-0. PMID 37496001